CLINICAL TRIAL: NCT04501211
Title: Open Label Transdermal Granisetron to Relieve Chronic Nausea and Emesis and to Reduce Medical Utilization in Patients With Gastroparesis
Brief Title: Open Label Transdermal Granisetron to Relieve Chronic Nausea and Emesis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Abandoned due to limited resources
Sponsor: Indiana University (Other)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Principal Investigator, John M. Wo, Professor of Gastroenterology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1706966663
Record Dates: First submitted 2018-10-31; First posted 2020-08-06 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patch arm (Other): Transdermal Granisetron patch to be given for application for 24 weeks with 2 weeks on and one week off pattern for a total of 24 weeks
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Granisetron — transdermal sancuso patch
  Other Names: sancuso patch

SUMMARY:
To determine the efficacy of open -label transdermal patch on chronic nausea and emesis in patients with gastroparesis

DETAILED DESCRIPTION:
Gastroparesis is a chronic syndrome associated with a delay in stomach emptying. The clinical presentation of gastroparesis is very heterogeneous but can generally categorized into emesis-predominant, regurgitation-predominant and dyspeptic-predominant gastroparesis.

The underlying cause of nausea is very difficult to identify, and physician is often treat nausea symptomatically with anti-nausea and anti-emetic medications.4, 5 Phenothiazine's such as prochlorperazine (Compazine®), promethazine (Phenergan®), and trimethobenzamide (Tigan®) have significant side effects and the potential of withdraw symptoms when these medications are stopped. Serotonin (5- HT3) antagonists have central emetic effects and have been utilized in acute chemotherapy-induced nausea and vomiting. Ondansetron, granisetron, palonosetron, and dolasetron are currently available as 5- HT3 antagonists for nausea and emesis. Oral dissolving and oral tablet formulation is suboptimal in outpatients with frequent emesis. Transdermal formulation may be optimal for patients with prolong nausea and vomiting, but data for chronic symptoms associated with gastroparesis is very limited.

An open-label, uncontrolled treatment pilot study with 2-week cycles of granisetron transdermal patch for 24 weeks in patients with chronic nausea and vomiting associated with gastroparesis

ELIGIBILITY:
Inclusion Criteria:

1. Documented delayed gastric emptying by 4-hr gastric scintigraphy using the standard protocol within 12 months.6
2. Symptoms of gastroparesis for >3 months
3. No upper gastrointestinal obstruction by upper endoscopy, barium radiograph, or CT scan.
4. Gastroparesis Cardinal Symptom Index Nausea-Vomiting (GCSI-N/V) subscale score of >2.0 during a 2-week run-in period.

Exclusion Criteria:

* 1. Baseline ECG with QTc >450ms in men or >470ms in women 2. Prolong QT syndrome 3. History of Torsade's de pointes, ventricular tachycardia, cardiomyopathy or implanted cardiac defibrillator 4. Use of cardiovascular antiarrhythmic medications 5. Strong CYP1A1 and CYP3A4 inhibitors that will inhibit metabolism of 5-HT3 antagonists

  1. CYP1A1 Inhibitors: pifithrin, ethinyl estradiol, fluvoxamine (Luvox®), mexiletine, miconazole, oltipraz , perazine, rofecoxib, aminobenzotriazole, isoniazid, lidocaine, zileuton (Zyflo®)
  2. CYP3A strong inhibitors: boceprevir, cobicistat (Tybost®), conivaptan (Vaprisol®), danoprevir and ritonavir, elvitegravir and ritonavir, grapefruit juice, indinavir and ritonavir, itraconazole (Onmel®, Sporanox®), ketoconazole, lopinavir and ritonavir (Kaletra®), paritaprevir and ritonavir and (ombitasvir and/or dasabuvir), posaconazole (Noxafil®), ritonavir (Norvir®), saquinavir and ritonavir), tipranavir and ritonavir, troleandomycin, voriconazole (Vfend®), clarithromycin (Biaxin®), diltiazem (Cardizem®, Cartia®, Dilacor®, Dilt-CD®, Diltia XT®, Taztia XT®, Tiazac®), idelalisib (Zydelig®), nefazodone (Serzone®), nelfinavir (Viracept®) 6. Serotonergic drugs that may increase the risk of serotonin syndrome

  <!-- -->

  1. Selective serotonin reuptake inhibitors (SSRIs)
  2. Selective norepinephrine reuptake inhibitors (SNRIs)
  3. Others: monoamine oxidase inhibitors: selegiline (Emsam®), isocarboxazid (Marplan®), pheneizine (Nardil®), tranylcypromine (Parnate®), mirtazapine (Remeron®), fentanyl (Sublimaze®), lithium (Eskalith®, Lithobid®), tramadol (ConZip®, Rybix®, Ryzolt®, Ultram®), intravenous methylene blue 7. Any comorbid condition that may prohibit enrollment 8. Other causes of nausea identified by the investigators other than gastroparesis 9. Any contraindications for 5HT3 receptor antagonists 10. Non-ambulatory patients: bed-ridden, nursing home resident, etc. 11. Pregnancy 12. Unable to give own informed consent 13. Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improvement in chronic nausea and emesis. | 24 weeks
  Incidence of participants who benefitted from the use of the patch at the end of 2 weeks, 8 weeks, 16 weeks and 24 weeks as assessed by the Gastroparesis Cardinal Symptom Index Nausea-Vomiting (GCSI-N/V). Mean subscale scores will compared for improvement every 6 weeks.

SECONDARY OUTCOMES:
Number of participants with reduced medical utilization for gastroparesis. | 24 weeks
  Incidence of participants who required less medical resources during treatment by comparing subject self-reports of medication usage, ER visits, home health therapy, and hospitalizations 12 weeks before, 12 weeks after, and 24 weeks after treatment with open label transdermal granisetron.

CONTACTS AND LOCATIONS:
Overall Officials: John M Wo, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No